CLINICAL TRIAL: NCT05047523
Title: A Multicenter, Randomized, Controlled, Open-label, Rater-blinded Study to Evaluate Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of ALXN1840 Versus Standard of Care in Pediatric Participants With Wilson Disease
Brief Title: Study of ALXN1840 Versus Standard of Care in Pediatric Participants With Wilson Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to terminate the program
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALXN1840-WD-302; 2021-001015-82 (EudraCT Number)
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Wilson Disease
Keywords: Wilson Disease; Pediatric
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is rater-blinded for the Unified Wilson Disease Rating Scale (UWDRS) assessment only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALXN1840 (Experimental): ALXN1840 will be administered at one of two starting doses, with incremental dose increases permitted.
  Interventions: Drug: ALXN1840
- Standard of Care (Active Comparator): Participants will receive their current therapy or initiate Standard of Care therapy.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: ALXN1840 — Administered as an oral tablet.
  Other Names: Formerly WTX101
  Arms: ALXN1840
Drug: Standard of Care — Depending on the site/region, participants randomized to receive Standard of Care treatment will receive trientine, penicillamine, zinc, or a combination of these medicines, administered according to standard regimens.
  Arms: Standard of Care

SUMMARY:
This study is being conducted to evaluate the efficacy, safety, pharmacokinetics (PK), and pharmacodynamics of ALXN1840 versus standard of care in pediatric participants with Wilson disease (WD).

DETAILED DESCRIPTION:
Participants who complete the 48 weeks of treatment in Period 1 will have the option to receive ALXN1840 for 24 weeks in Period 2 (open-label extension).

Safety will be monitored throughout the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of Wilson Disease by Leipzig Score ≥ 4.
2. Adequate venous access to allow collection of required blood samples.
3. Able to swallow intact ALXN1840 tablets or mini-tablets.
4. Willing to avoid intake of foods and drinks with high contents of copper.
5. Willing and able to follow protocol-specified contraception requirements.

Key Exclusion Criteria:

1. Decompensated hepatic cirrhosis or MELD score > 13 (ages 12 to <18) or PELD score > 13 (ages 3 to < 12).
2. Modified Nazer score > 7.
3. Clinically significant gastrointestinal bleed within past 3 months.
4. Alanine aminotransferase (ALT) > 2 × upper limit of normal (ULN) for participants treated for > 28 days with WD therapy or ALT > 5 × ULN for treatment-naïve participants or participants who have been treated for ≤ 28 days.
5. Marked neurological disease requiring either nasogastric feeding tube or intensive inpatient medical care.
6. Hemoglobin less than lower limit of the reference range for age and sex.
7. History of seizure activity within 6 months prior to informed consent/assent.
8. Participants in renal failure, defined as in end-stage renal disease on dialysis (chronic kidney disease stage 5) or estimated glomerular filtration rate < 30 milliliters/minute/1.73 meter squared.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S. Swenson, MD, PhD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (18):
- Australia (2):
  - Research Site, Parkville
  - Research Site, South Brisbane
- France (2):
  - Research Site, Lille
  - Research Site, Toulouse
- Germany (2):
  - Research Site, Hanover
  - Research Site, Tübingen
- Japan (4):
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Meguro-ku
  - Research Site, Sapporo
- Research Site, Warsaw, Poland
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Esplugues de Llobregat
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1840-WD-302&attachmentIdentifier=89039cf8-1563-49de-8885-40fcb43b5b3b&fileName=alxn1840-wd-302-CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 2 periods: Primary Evaluation Period (PEP) and Open-label Extension (OLE) Period. Participants who completed the 48-week PEP were offered the opportunity to continue treatment in an up to 24-week OLE Period.
Pre-assignment Details: Per prespecified analysis, participants were randomized, stratified by cohort, in 1:1 ratio to ALXN1840 or continued treatment with Standard of Care (SoC) in Cohort 1 or as continued or initial therapy in Cohort 2 for the PEP. The stratification was not applicable to the OLE Period. Data was collected for the OLE Period by dose received irrespective of the cohort assigned during randomization.
Groups:
- Cohort 1: ALXN1840: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) received titrated doses of ALXN1840 orally for up to 48 weeks in the PEP.
- Cohort 1: SoC Therapy: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) continued to receive SoC therapy according to the local package label for up to 48 weeks in the PEP.
- Cohort 2: ALXN1840: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received titrated doses of ALXN1840 orally for up to 48 weeks in the PEP.
- Cohort 2: SoC Therapy: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received SoC therapy according to the local package label for up to 48 weeks in the PEP.
- ALXN1840/ALXN1840: Participants who were randomized to the ALXN1840 group during the PEP and who completed the 48-week PEP were offered the opportunity to participate in the OLE Period and continued to receive ALXN1840 for up to 24 additional weeks.
- SoC Therapy/ALXN1840: Participants who were randomized to the SoC group during the PEP and who completed the 48-week PEP were offered the opportunity to participate in the OLE Period and received ALXN1840 for up to 24 additional weeks.
Period: Primary Evaluation Period (48 Weeks)
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy | ALXN1840/ALXN1840 | SoC Therapy/ALXN1840
Started | 15 | 16 | 4 | 5 | 0 | 0
Received at Least 1 Dose of Study Drug | 15 | 16 | 4 | 5 | 0 | 0
Completed | 12 | 11 | 0 | 1 | 0 | 0
Not Completed | 3 | 5 | 4 | 4 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 2 | 4 | 3 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Extension Period (24 Weeks)
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy | ALXN1840/ALXN1840 | SoC Therapy/ALXN1840
Started | 0 | 0 | 0 | 0 | 12 | 12
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 12 | 12
Completed | 0 | 0 | 0 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 9 | 9
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 8 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of ALXN1840 or SoC treatment.
Groups:
- Cohort 1: ALXN1840: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) received titrated doses of ALXN1840 orally for up to 48 weeks in PEP.
- Cohort 1: SoC Therapy: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) continued to receive SoC therapy according to the local package label for up to 48 weeks in PEP.
- Cohort 2: ALXN1840: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received titrated doses of ALXN1840 orally for up to 48 weeks in PEP.
- Cohort 2: SoC Therapy: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received SoC therapy according to the local package label for up to 48 weeks in PEP.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy | Total
Number analyzed (Participants) | 15 | 16 | 4 | 5 | 40
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 6 | 6 | 3 | 3 | 18
  Adolescents (12-17 years) | 9 | 10 | 1 | 2 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 3 | 15
  Male | 10 | 12 | 1 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 0 | 0 | 9
  Not Hispanic or Latino | 10 | 11 | 4 | 5 | 30
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 1 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 9 | 9 | 0 | 2 | 20
  More than one race | 1 | 0 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 48 in Non-ceruloplasmin-bound Copper in Plasma
Description: Plasma samples were planned to be collected to measure ceruloplasmin-bound copper. Due to the early termination of the study, data for this Outcome Measure were not collected for any of the cohorts.
Time Frame: Baseline, Week 48
Population: FAS included all participants who received at least 1 dose of ALXN1840 or SoC treatment. Due to the early termination of the study, data for this Outcome Measure were not collected for any of the cohorts.
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Primary Evaluation Period
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered the study drug and which did not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs with onset after the first dose of study intervention or existing events that worsened in severity after the first dose of study intervention. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who received at least 1 dose of ALXN1840 or SoC treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 15 | 16 | 4 | 5
Participants | 13 | 13 | 3 | 4

3. Secondary Outcome: Area Under the Effect Versus Time Curve (AUEC) for Plasma Total Copper and Direct NCC
Time Frame: Week 48
Population: Pharmacodynamic (PD) analysis set included all participants who had sufficient plasma samples to enable the calculation of pharmacokinetic (PK) parameters and provide PK/PD profiles. Here, 'Overall number of participants analyzed' = participants evaluable for this Outcome Measure. No participants were evaluable for this Outcome Measure for Cohort 2: ALXN1840.
Measure: Mean (Standard Deviation); unit: nanograms (ng)*hours (hr)/milliliter(mL)
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 11 | 11 | 0 | 1
nanograms (ng)*hours (hr)/milliliter(mL)
  Total Copper | 6342.909 (3038.3317) | 7528.864 (4167.2110) |  | 16369.000 (NA) — Data could not be calculated due to single participant.
  Direct NCC | 3882.473 (1716.4565) | 3067.864 (1524.9183) |  | 4214.000 (NA) — Data could not be calculated due to single participant.

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of ALXN1840 for Plasma Total Molybdenum and Plasma Ultrafiltrate Molybdenum Concentrations
Time Frame: Week 48
Population: PK analysis set included all participants who had sufficient plasma samples to enable the calculation of PK parameters and provide PK/PD profiles. Here, 'Overall number of participants analyzed' = participants evaluable for this Outcome Measure. No participants were evaluable for this Outcome Measure for Cohort 2: ALXN1840.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 12 | 11 | 0 | 1
ng/mL
  Plasma Total Molybdenum | 183.150 (110.4736) | 209.355 (114.3741) |  | 307.000 (NA) — Data could not be calculated due to single participant.
  Plasma Ultrafiltrate Molybdenum | 13.733 (8.6186) | 17.708 (27.9548) |  | 9.910 (NA) — Data could not be calculated due to single participant.

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the End of the Dosing Interval (AUCtau) of ALXN1840 for Plasma Total Molybdenum and Plasma Ultrafiltrate Molybdenum
Time Frame: Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 11 | 11 | 0 | 1
ng*hr/mL
  Plasma Total Molybdenum | 4498.082 (3054.8300) | 2931.045 (1694.3512) |  | 4261.100 (NA) — Data could not be calculated due to single participant.
  Plasma Ultrafiltrate Molybdenum | 233.154 (145.7960) | 144.627 (88.6710) |  | 129.370 (NA) — Data could not be calculated due to single participant.

ADVERSE EVENTS:
Time Frame: Baseline up to Week 76
Description: Safety analysis set included all participants who received at least 1 dose of ALXN1840 or SoC treatment.
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy | ALXN1840/ALXN1840 | SoC Therapy/ALXN1840
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/4 | 0/5 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/16 | 0/4 | 0/5 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 13/15 | 12/16 | 2/4 | 4/5 | 6/12 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ALXN1840 (N=15) | Cohort 1: SoC Therapy (N=16) | Cohort 2: ALXN1840 (N=4) | Cohort 2: SoC Therapy (N=5) | ALXN1840/ALXN1840 (N=12) | SoC Therapy/ALXN1840 (N=12)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ALXN1840 (N=15) | Cohort 1: SoC Therapy (N=16) | Cohort 2: ALXN1840 (N=4) | Cohort 2: SoC Therapy (N=5) | ALXN1840/ALXN1840 (N=12) | SoC Therapy/ALXN1840 (N=12)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 4 (5)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (7) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early termination of the study, data for the efficacy endpoints were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT05047523/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT05047523/SAP_001.pdf